CLINICAL TRIAL: NCT06251440
Title: Transabdominal Fetal Reduction in Higher Order Multiple Pregnancies - a Pioneer Study in Nepal
Brief Title: Initial Experience of Transabdominal Fetal Reduction in Nepal
Status: Completed | Type: Observational
Sponsor: Grande International Hospital, Nepal (Other)
Responsible Party: Principal Investigator, PRAJWAL DAHAL, Principal Investigator, Grande International Hospital, Nepal
Other Study IDs: 20/2020
Record Dates: First submitted 2024-01-31; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: In Vitro Fertilization
Keywords: Fetal reduction; Multifetal gestation; In Vitro fertilization
MeSH Terms: interventions — Pregnancy Reduction, Multifetal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Fetal Reduction — Under ultrasound guidance, intracardiac injection of 0.2 to 3.0 ml of 15% weight/volume (2 miliequivalent/mililiter ) potassium chloride (KCl) was administered via transabdominal route
  Other Names: Selective fetal reduction

SUMMARY:
Multifetal pregnancies are common in in vitro fertilization. Multifetal gestation increases maternal and fetal morbidity and mortality. We perform fetal reduction in our hospital by intra-thoracic injection of potassium chloride. This manuscript is description of our initial experience.

DETAILED DESCRIPTION:
Assisted reproductive technology and stimulated conception have led to an increase in the prevalence of high order multifetal pregnancies (MFPs) in recent times. MFPs are associated with high maternal and fetal complications. Fetal mortality and morbidity are due to complications of prematurity. Prevalence of pregnancy induced hypertension, pre-eclampsia, eclampsia, antepartum hemorrhage, post-partum hemorrhage, gestational diabetes and difficult deliveries are more in mother with MFP. Embryo/Fetal reduction in high order MFPs helps in prolongation of gestation. Multifetal pregnancy reduction (MFPR) is secondary prevention of the risks associated with MFP. Trans-abdominal intracardiac injection of KCl is a simple, safe and effective technique for MFPR. We are among the first few centers in Nepal doing MFPR. In this study, we are sharing our initial experience of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* pregnant females with multifetal gestation who opt to undergo fetal reduction

Exclusion Criteria:

* who do not give consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females with multiple pregnancy
Study Population: Multifetal pregnancies referred from the obstetrics and gynecology department of our hospital, different other hospitals and in vitro fertilization (IVF) centers across the country underwent ultrasound-guided transabdominal embryo/ fetal reduction procedure between February 2018 to April 2023 in our department.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Transabdominal ultrasonography guided fetal reduction is safe and effective in first trimester | 4.5 years
  To share initial experience of transabdominal multifetal pregnancy reduction (MFPR) in Nepal

CONTACTS AND LOCATIONS:
Overall Officials: Sharma Poudel, MD, Principal Investigator — Grande International Hospital
Locations (1):
- Prajwal Dahal, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No